CLINICAL TRIAL: NCT04022447
Title: Dupilumab Effectiveness in Severe Asthma: a Cohort Study From a Nationwide Early Access
Brief Title: Dupilumab for Severe Asthma in a Real Life Setting
Acronym: DUPI-France
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HAO 18053
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Severe Asthma
Keywords: dupilumab; asthma; real life; safety
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dupilumab — retrospective data collection
  Other Names: retrospective non interventional

SUMMARY:
Dupilumab is a monoclonal anti-IL-4/13Rα antibody developed for severe asthma (SA). In France, mepolizumab was commercialized in February 2018. Before this date, many SA patients had reached a therapeutic dead end, with uncontrolled disease despite maximal available treatment. Upon the request of lung specialists involved in SA, French health authorities approved an early access program (temporary Use Authorization) allowing early access to dupilumab (before EMA's decision) from September 2017 to January 2018, for SA patients demonstrating unacceptable steroids side effects and/or life-threatening exacerbations, irrespective of their T2 status.The aim of this retrospective study was to describe the characteristics of SA patients included in the early access program and to assess changes in asthma control after a 12 months treatment.

DETAILED DESCRIPTION:
Introduction:

Asthma is a worldwide burden affecting more than 300 millions patients. Although the vast majority of asthma patients suffer from mild to moderate diseases whose symptoms can be assessed with inhaled corticosteroids (CSI) and bronchodilators, 3.7% of them present with severe asthma (SA). SA is defined as an asthma remaining uncontrolled despite adherence with maximal optimized therapy and treatment of contributory factors, or that worsens when high dose treatment is decreased. SA represents a small proportion of patients but the very heart of the asthma problem with tremendous health costs, high morbidity and significant mortality. Thus it has been the center of therapeutic research interest for the past decade and different treatments have achieved development and reglementary approvals. Among them, dupilumab is a fully human monoclonal antibody targeting the alpha subunit of the interleukin 4 receptor, blocking both IL-4 and IL -13 pathways. It is therefore interacting with the type 2 inflammation response observed in eosinophilic asthma. The French Ministry of Health therefore opened a window of appeals for TUA from September 2017 to January 2018, allowing early access to dupilumab for SA patients demonstrating unacceptable steroids side effects and/or life-threatening exacerbations, irrespective of their T2 status. By that time indeed, phase 3 randomized clinical trials (RCT) on eosinophilic patients had not yet been published.

In this phase IV real-life study with no placebo group, the investigators aimed to describe patients' characteristics and to evaluate the efficacy and safety of Dupilumab on non-selected SA patients.

Method:

This multicenter retrospective observational real-life study was conducted at 13 public teaching hospitals across the country. All French SA patients who received dupilumab under the TUA between September 2017 and January 2018 were included in the survey, as long as they had received at least one injection and completed at least one follow-up visit in the first 12 months of treatment. No inclusion criteria were required, but patients' files had previously been screened through by health authorities and validated by Sanofi to allow dupilumab TUA. Physicians had had to certify that patients had SA with no other treatment available at that time, and that poor asthma control and/or severe steroid side effects required scaling up treatment. Patients were not required to have eosinophilia. However, patients were excluded from the TUA if they presented with previous hypereosinophilia > 1500/mm3, as symptomatic hypereosinophilia has previously been described with dupilumab in this particular population.

Investigators were free to decide on the frequency of visits, blood tests and function assessments, as to define the tools of control assessment, in adequacy with their usual practice. On line and paper questionnaires were retrospectively filled.

Main objective of the study was to describe asthma control at 12 months and secondary objectives were descriptive data of the population, efficacy, safety and tolerability of dupilumab treatment. Statistics of patients' characteristics were compiled. Efficacy was assessed in the per-protocol population, defined as all the patients who completed visits at 3, 6 and/or 12 months. Differences between baseline and follow-up visits were compared by Wilcoxon signed-rank test and rank-sum test. ACT evolution during study was assessed with a mixed linear model.

Response was eventually assessed by each investigator using the GETE score (5 categories, graded from 1 to 5, respectively defining the disease control as excellent - good - moderate - poor and worsening). Categories 1 and 2 are considered as good response.

Clinical response was defined as gain of ACT score of more than 5 points compared to previous assessment or ACT > 18. Time to first clinical response was evaluated using Kaplan-Meier curves.

Safety and tolerability were evaluated on the basis of each investigator notifications The protocol was approved by the institutional review boards of the French learned society for respiratory medicine - Société de Pneumologie de Langue Française and of the Paris University Hospitals - Assistance Publique - Hôpitaux de Paris. The independent Committee for the protection of persons (CPP) gave a favourable opinion. All patients provided oral consent to the collection of their data. As a non interventional retrospective study, no written consent was required.

ELIGIBILITY:
Inclusion Criteria:

* French patient with Severe Asthma
* Administration of dupilumab under the TUA between September 2017 and January 2018, with at least one injection
* Realization of at least one follow-up visit in the first 12 months of treatment

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between September 2017 and January 2018, 86 TUA applications were registered from 13 different teaching hospitals nationwide.
  17 patients did not eventually receive the treatment and 69 were thus screened for study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
asthma control with dupilumab | 12 months
  asthma control evaluated by Asthma Control Test
number of asthma exacerbations | 12 months
  number of self reported asthma exacerbations, defined by the use of oral steroids for at least 3 days
number of asthma-related hospitalizations | 12 months
  number of self reported or documented in the medical file asthma-related hospitalizations
FEV1 (Forced Expiratory Volume in 1 sec) | 12 months
  FEV1 (Forced Expiratory Volume in 1 sec) expressed in ml
oral steroids consumption | 12 months
  daily dose of prednisone (mg)

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAILLE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat-Claude Bernard University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dupin C, Belhadi D, Guilleminault L, Gamez AS, Berger P, De Blay F, Bonniaud P, Leroyer C, Mahay G, Girodet PO, Raherison C, Fry S, Le Bourdelles G, Proust A, Rosencher L, Garcia G, Bourdin A, Chenivesse C, Didier A, Couffignal C, Taille C. Effectiveness and safety of dupilumab for the treatment of severe asthma in a real-life French multi-centre adult cohort. Clin Exp Allergy. 2020 Jul;50(7):789-798. doi: 10.1111/cea.13614. Epub 2020 May 29. PMID 32469092